CLINICAL TRIAL: NCT05401773
Title: α-synuclein Seeding Activity in the Olfactory Mucosa in COVID-19 - A Pilot Study
Brief Title: α-synuclein Seeding Activity in the Olfactory Mucosa in COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1448/2020
Record Dates: First submitted 2022-06-01; First posted 2022-06-02 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- COVID-19 patients with olfactory dysfunction (Experimental): COVID-19 patients with olfactory dysfunction
  Interventions: Other: Real-time Quaking-Induced Conversion (RT-QuIC)
- COVID-19 patients without olfactory dysfunction (Experimental): COVID-19 patients without olfactory dysfunction
  Interventions: Other: Real-time Quaking-Induced Conversion (RT-QuIC)
- Healthy controls (Experimental): Healthy controls
  Interventions: Other: Real-time Quaking-Induced Conversion (RT-QuIC)
- Patients with Parkinson's disease (Experimental): Patients with Parkinson's disease
  Interventions: Other: Real-time Quaking-Induced Conversion (RT-QuIC)

INTERVENTIONS:
Other: Real-time Quaking-Induced Conversion (RT-QuIC) — RT-QuIC is increasingly used as diagnostic tools in synucleinopathies and has shown high sensitivity and specificity for the detection of α-synuclein seeds in CSF and tissue samples, including the olfactory mucosa in different patients' cohorts including Parkinson's patientients, patients with REM sleep behavior disorder (RBD), and patients with dementia with Lewy bodies.

SUMMARY:
Loss of the sense of smell is a characteristic feature of COVID-19 and likely related to viral invasion of the olfactory mucosa but is also a prodromal feature of PD. This constellation has kindled concerns that COVID-19 - similar to the Spanish Flu Pandemic in 1918 - might trigger a second wave of post-infectious parkinsonism. The main objective of the study is to probe for the presence of pathological α-synuclein assemblies in the olfactory mucosa of patients with COVID-19.

DETAILED DESCRIPTION:
Deposits of misfolded proteins are the cause of frequent neurological diseases such as Alzheimer's or Parkinson's disease. In Parkinson's disease, the misfolded protein alpha-synuclein is found in the olfactory mucosa of the nose, which contains nerve cells responsible for smell perception, from which the misfolded alpha-synuclein spreads further into the brain. The mechanisms that lead to this misfolding and the resulting damage to the nervous system are still unclear. One hypothesis is that inflammatory processes such as viral infections trigger the misfolding of alpha-synuclein in Parkinson's disease and can lead to its deposition. Based on this assumption and the striking involvement of the sense of smell in SARS-CoV-2 infection (COVID-19), the aim of this study is to investigate the olfactory epithelium of the nasal mucosa of COVID-19 patients for possible alpha-synuclein deposits by using nasal swabs.

We hypothesize that the invasion of olfactory neurons and subsequent inflammatory responses could trigger α-synuclein misfolding and aggregation. Therefore, we aim to investigate for the presence of α-synuclein seeding activity in the olfactory mucosa of subjects who have recovered from COVID-19 by using Real-time Quaking-Induced Conversion (RT-QuIC).

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be 18 years or older;
2. Participants are able to understand the aim of the study and the planned procedures;
3. Written informed consent form;
4. Participants fulfilling the criteria for one of the following groups:

   1. COVID-19 patients with OD:

      * Prior history of COVID-19 (clinical documentation plus corresponding positive PCR test) at least 3 months ago;
      * OD (Sniffin' sticks discrimination and identification both <13/16 items correct) persisting for at least 3 months after SARS-CoV-2 infection;
      * Negative antigen test on day of study inclusion;
      * No evidence of structural nasal pathologies possibly responsible for OD.
   2. COVID-19 patients without OD:

      * Prior history of COVID-19 (clinical documentation plus corresponding positive PCR test) at least 3 months ago;
      * No history of/current OD (Sniffin' sticks discrimination and identification both >12/16 items correct);
      * Negative antigen test on day of study inclusion.
   3. Healthy Controls:

      * No history of COVID-19 and negative SARS-CoV-2 antibody test unless subject is vaccinated;
      * Negative antigen test on day of study inclusion;
      * No history of OD;
      * Subjective and objective normal olfactory function (Sniffin' sticks discrimination and identification both >12/16 items correct). 10 Application for Clinical Research
   4. Patients with Parkinson's disease (n = 50):

      * Confirmed diagnosis of PD according to diagnostic criteria.
      * No history of COVID-19 and negative SARS-CoV-2 antibody test unless subject is vaccinated;
      * Negative antigen test on day of study inclusion;

Exclusion Criteria:

1. Patients:

   * History of OD prior to SARS-CoV-2 infection;
   * Pre-existent relevant neurological disorder;
   * Positive SARS-CoV-2 antigen test on day of study inclusion;
   * Patients with OD only: structural pathology possibly responsible for OD.
2. Healthy controls:

   * Pre-existent relevant neurological disorder;
   * History of/presence of olfactory dysfunction (Sniffin' sticks discrimination and identification both <13/16 items correct);
   * Positive SARS-CoV-2 antigen test on day of study inclusion;
   * Positive SARS-CoV-2 antibody test unless subject is vaccinated.
3. Patients with Parkinson's disease:

   * History of COVID-19;
   * Positive SARS-CoV-2 antigen test on day of study inclusion;
   * Positive SARS-CoV-2 antibody test unless subject is vaccinated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Demonstration of ⍺-synuclein seeding activity in the OM (assessed by RT-QuIC) in subjects who recovered from COVID-19 compared to healthy controls. | 2 years
  detection ⍺-synuclein seeding activity in olfactory mucosa of different patient groups

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Heim, MD PhD, Study Chair — Medical University Innsbruck
Locations (1):
- Medical University of Innsbruck, Innsbruck, Austria